CLINICAL TRIAL: NCT07231068
Title: A Dose-escalation and Dose-expansion Phase I/Phase II Clinical Study on the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of Dositinib Mesylate Tablets (90-1408) in the Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer With Positive EGFR Mutations
Brief Title: A Dose-escalation and Dose-expansion Phase I/Phase II Clinical Study of Dositinib Mesylate Tablets (90-1408) in the Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer With Positive EGFR Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YD-Dox-200511
Record Dates: First submitted 2025-09-24; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; EGFR mutation; Dositinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Dose-escalation part and dose-expansion part
  Interventions: Drug: Dositinib mesylate tablets

INTERVENTIONS:
Drug: Dositinib mesylate tablets — Dose-escalation part: Subjects received 90-1408 at doses of 20, 40, 80, 160, 200 and 240 mg. A single oral dose was administered on Cycle 1 Day 1, then once daily from Day 8 onward. Dosing occurred in the morning, with 21 days of continuous treatment per cycle.
  Dose-expansion part: Subjects received 90-1408 orally at a dose of 80, 160 and 200 mg, administered once daily for 21 consecutive days per cycle.
  Other Names: 90-1408

SUMMARY:
This is an open label phase I/phase II clinical study designed to evaluate the safety, tolerability, pharmacokinetics, preliminary efficacy of Dositinib in participants of locally advanced or metastatic non-small cell lung cancer with positive EGFR mutation.

DETAILED DESCRIPTION:
Dositinib is an EGFR-TKI. There are two parts in the study. Phase I is dose escalation study, and Phase II is dose expansion study. Phase I will be conducted using 3+3 dose escalation method. In Phase II, 3 dose levels will be chosen to further evaluate the safety and efficacy of Dositinib.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old (including 18 and 75 years old), male or female.
2. Histologically or cytologically confirmed patients with locally advanced NSCLC (stage IIIB / IIIc) or metastatic NSCLC (stage IV) who are unable to undergo radical surgery or radiotherapy (International Alliance against cancer, 8th Edition, 2017).
3. Locally advanced or metastatic NSCLC patients who have documentation of disease progression (with imaging evidence) while on previous continuous treatments with EGFR-TKI (such as gefitinib, erlotinib, icotinib, afatinib, etc., excluding the third-generation EGFR TKI drugs), or cannot tolerate the treatments for various reasons (only applicable to dose escalation part).
4. Patients with confirmed EGFR activating mutations that are sensitive to EGFR TKI at any time after initial diagnosis, in dose escalation part including G719X, exon 19 deletion, L858R, L861Q, in dose expansion part including exon 19 deletion and L858R.
5. No prior systemic antitumor therapy for locally advanced or metastatic NSCLC (patients who have received first-line chemotherapy but not TKI treatment can be enrolled). Patients who have undergone radical surgery, radical chemoradiotherapy or adjuvant treatment (chemotherapy, radiotherapy) for early-stage NSCLC and have experienced disease recurrence or metastasis later can be enrolled (only applicable to dose expansion part).
6. According to RECIST 1.1 response evaluation criteria in solid tumours, the patient has at least one imaging (CT, MRI) measurable or evaluable lesion, and accurate and repeatable measurement can be made at baseline, such as CT or MRI. In the dose expansion part, for the 160 mg and 200 mg dose groups, at least one measurable intracranial lesion is required in 20 to 30 patients with brain metastases. The long diameter of the lesion is more than or equal to 10 mm (if the lesion is a metastatic lymph node, the short diameter is more than or equal to 15 mm), and the lesion has not received radiotherapy or biopsy in the past (if the patient has only one target lesion and needs biopsy, the target lesion can be biopsied, and the time interval between the biopsy and the baseline assessment of the tumor in the screening period must be more than 2 weeks, and the target lesion still meets the definition in RECIST1.1 after biopsy). The same test method should be used in the follow-up evaluations.
7. Subjects with ECOG performance score of 0-1.
8. Patients whose life expectancy is at least 12 weeks.
9. Patients have adequate important organ functions during screening, including: a. The absolute neutrophil count (NEUT#) ≥ 1.5 x 10^9/L without using hematopoietic stimulating factor within 14 days before the first administration; b. Platelet count ≥ 100 x 10^9 / L without using hematopoietic stimulating factor or blood transfusion within 14 days before the first administration; c. Hemoglobin>90g/L without using hematopoietic stimulating factor or blood transfusion within 14 days before the first administration; d. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN (ULN = upper limit of normal value) or ≤ 5 x ULN (patients with hepatic metastases); e. Total bilirubin ≤1.5 x ULN (ULN = upper limit of normal value) or ≤ 3 x ULN (patients with hepatic metastase); f. Coagulation function INR ≤ 1.5; g. Serum creatinine ≤ 1.5 x ULN (ULN = upper limit of normal value) and creatinine clearance rate (calculated by Cockcroft and Gault formula) ≥ 50ml / min.
10. Female subjects of childbearing age must confirm that the blood pregnancy test is negative and agree to use effective contraceptive measures during the use of the study drug and within 90 days after the last administration.

    In this program, female subjects of childbearing age are defined as sexually mature women. (1) No hysterectomy or bilateral oophorectomy is performed; (2) Natural amenorrhea doesn't last for 12 consecutive months (amenorrhea after cancer treatment does not exclude fertility) (i.e., menstruation occurred at any time in the previous 12 consecutive months); if the female partner of a male subject is fertile, the subject must agree to take adequate contraceptive measures from the first administration of the study treatment to 90 days after the last administration of the study treatment.
11. The subjects should give informed consent to the study and sign the informed consent form before the trial.

Exclusion Criteria:

1. Within 28 days before the first administration of the study treatment, the patients have used any chemotherapy drugs and / or immunotherapy drugs in the previous treatment regimen or clinical study; or have undergone major surgery (excluding vascular access establishment surgery) or received > 30Gy within 28 days before the first administration of the study treatment. In addition to the local palliative radiotherapy for bone metastases, the patient have used an experimental drug or other anticancer drugs in the previous treatment regimen or clinical study within 14 days before the first administration of the study treatment, or stopped using other experimental drugs or anticancer drugs for less than 5 ×half-life (e.g., erlotinib less than 8 days, gefitinib less than 10 days, icotinib less than 2 days, afatinib less than 8 days).
2. Patients who have used the third generation EGFR TKI drugs (such as Osimertinib, rociletinib (co-1686), olmutinib (hm61713), asp8273, egf816, Mefatinib, Avitinib, etc.).
3. Patients who participated in other therapeutic clinical trials within one month before the first administration (patients who discontinue the experimental drug after more than five half-lives of the drug can be included in the study).
4. The patients are using (or cannot stop using) CYP3A4 strong inhibitor or inducer or Chinese herbal medicine with anti-tumor indications.
5. Patients who did not recover from the adverse events caused by previous anti-tumor therapy (recovered to ≤ 1 grade) (except for alopecia).
6. Patients with other malignant tumors within 5 years before the start of treatment (except for basal cell carcinoma or squamous cell carcinoma of the skin that is not melanoma, breast / cervical carcinoma in situ, superficial bladder carcinoma and other carcinoma in situ who have received radical treatment and no evidence of recurrence).
7. Any condition that affects the patients' swallowing of the drug and seriously affects the absorption or pharmacokinetic parameters of the investigational drug, including any kind of uncontrollable nausea and vomiting, chronic gastrointestinal diseases, inability of the patient to swallow the drug, history of gastrointestinal resection or surgery.
8. Patients with known organ transplantation.
9. Meet any of the following cardiac criteria: QTc interval > 450ms in male and > 470ms in female (QTc interval calculated by fridericia formula). All kinds of ECG morphological abnormalities with clinical significance, such as complete left bundle branch block, grade III block, grade II block, PR interval > 250ms. Various factors that may increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of immediate family members with long QT syndrome or unexplained sudden death before 40 years of age, and the use of any drug with known QT interval prolongation.
10. Past medical history: interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, active interstitial lung disease with clinical evidence; patients with active pulmonary tuberculosis (TB) who are receiving anti tuberculosis treatment or received anti tuberculosis treatment within one year before screening.
11. Pulmonary function test: forced expiratory volume in one second (FEV1) / forced vital capacity (FVC) < 70%, FEV1% < 30%, or DLCO% < 40%.
12. Patients with spinal cord compression, or meningeal metastasis, or symptomatic and untreated brain metastasis (except those who are asymptomatic, stable, and do not need steroid therapy for more than 4 weeks before the start of study treatment).
13. The patients have a history of hypersensitivity to the active ingredients or inactive excipients of the study drug, drugs with chemical structure similar to the study drug or similar drugs, etc.).
14. At any time after the initial diagnosis, there are confirmed EGFR 20 exon insertion mutations.
15. Subjects are in the stage of acute infection and need medical treatment.
16. In the active stage of hepatitis B or hepatitis C: HBsAg positive and HBV DNA ≥ 10^3 copies/mL or ≥ 200 IU/mL (HBV DNA is required when HBsAg is positive), HCVAb positive and HCV-RNA ≥ 10^3 copies/mL (HCV-RNA is required when HCVAb is positive).
17. Subjects are HIV positive.
18. Subjects with a clear history of mental disorders and who have taken medication for treatment
19. Subjects have a history of drug abuse.
20. Pregnant or lactating women.
21. Women of childbearing age and fertile men can not take effective contraceptive measures during the period from signing the informed consent to 90 days after the last use of the study drug.
22. The researcher believes that there are other factors that may affect the results of the study and interfere with the whole process of the study, including past or existing physical conditions, treatment or laboratory abnormalities, etc.; or the researcher believes that participating in the study can not maximize the benefits of the patients.
23. Subjects are not suitable to participate in this study for any reason in the judgment of the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | From enrollment to the end of the study, up to 28 days after the end of study treatment.
  AEs are assessed based on NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of 90-1408 in Single Administration | Up to 144 hours post-dose.
Pharmacokinetics (PK): Time to Maximum Plasma Concentration (Tmax) of 90-1408 in Single Administration | Up to 144 hours post-dose.
Pharmacokinetics (PK): Area Under the Plasma Concentration Curve (AUC) of 90-1408 in Single Administration | Up to 144 hours post-dose.
Pharmacokinetics (PK): Elimination Half-Life (t1/2) of 90-1408 in Single Administration | Up to 144 hours post-dose.
Pharmacokinetics (PK): Steady-State Valley Concentration (Css-min) of 90-1408 in Multiple Administration | Up to Day 29.
Pharmacokinetics (PK): Steady-State Peak Concentration (Css-max) of 90-1408 in Multiple Administration | Up to Day 29.
Pharmacokinetics (PK): Mean Steady-State Concentration (Css-ave) of 90-1408 in Multiple Administration | Up to Day 29.
Pharmacokinetics (PK): Elimination Half-Life (t1/2) of 90-1408 in Multiple Administration | Up to Day 29.
Effectiveness Evaluation: Overall Response Rate (ORR) | Up to approximately 60 months.
Effectiveness Evaluation: Duration of Response (DOR) | Up to approximately 60 months.
Effectiveness Evaluation: Disease Control Rate (DCR) | Up to approximately 60 months.
Effectiveness Evaluation: Progression-Free Survival (PFS) | Up to approximately 60 months.
Effectiveness Evaluation: Overall Survival (OS) | From enrollment until death from any cause, up to approximately 60 months.
Effectiveness Evaluation: Intracranial Progression-Free Survival (iPFS) | Up to approximately 60 months.
Effectiveness Evaluation: Intracranial Overall Response Rate (iORR) | Up to approximately 60 months.
Evaluation of Drug Metabolic Profiles: Metabolic Profiles of 90-1408 and Its Metabolites in Plasma and Urine | Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Junling Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Henan Provincial Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No